CLINICAL TRIAL: NCT03542266
Title: A Multi-center Phase II Study of CC486-CHOP in Patients With Previously Untreated Peripheral T-cell Lymphoma
Brief Title: CC486-CHOP in Patients With Previously Untreated Peripheral T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1711018777
Record Dates: First submitted 2018-05-18; First posted 2018-05-31 (Actual); Results first posted 2021-05-20 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-07

CONDITIONS: Previously Untreated Peripheral T-cell Lymphoma
Keywords: Peripheral T-cell Lymphoma; Azacitidine; Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma | interventions — Azacitidine

STUDY DESIGN:
Intervention Model Description: This is a phase II, multi-center study to determine the efficacy and safety of first-line CC-486 plus CHOP in patients with PTCL who have received no prior systemic therapy. The study has a sample size of 20, and follows two-stage minimax design for primary efficacy analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CC486 +CHOP (Experimental): CC486 +CHOP
  Interventions: Drug: CC-486 Administration; Drug: CHOP Administration

INTERVENTIONS:
Drug: CC-486 Administration — CC-486 at 300 mg once daily is to be administered Cycle 1, Day -6 to 0 and Cycles 1 to 5, Day 8 to 21. Antiemetic prophylaxis is recommended before dosing. All efforts should be made to administer CC-486 on all scheduled days of the Cycle 1 priming dosing (7 days, Cycle 1 Day -6 to Cycle 1 Day 0) and the Cycle 1-5 dosing (14 days, Day 8-21). A dose missed earlier in a day can be administered later that day as long as it is taken at least 8 hours before the next scheduled dose. Any missed dose should not be taken beyond the last scheduled day of CC-486 administration for the cycle, but should be returned by the subject for CC 486 accountability. If vomiting occurs after a dose of CC-486 is administrated, that dose should not be made up later that day.
  Other Names: Oral Azacitidine
Drug: CHOP Administration — CHOP is to be administered on Days 1 to 5 of Cycles 1-6. Chemotherapy can be administer within +72h or -24h of Day 1 of each scheduled Cycle. Preparation and infusion rate are according to the package insert and local practice. The doses to be used are:
  Cyclophosphamide: 750 mg/m2 IV on day 1 Doxorubicin: 50 mg/m2 IV on day 1 Vincristine: 1.4 mg/m2 IV (not to exceed 2.0 mg total) on day 1 Prednisone: 100 mg PO days 1-5

SUMMARY:
This is a phase II, multi-center study to determine the efficacy and safety of first-line CC-486 plus CHOP in patients with PTCL who have received no prior systemic therapy. The study has a sample size of 20, and follows two-stage minimax design for primary efficacy analysis.

DETAILED DESCRIPTION:
Study Summary:

This is a phase II, multi-center study to determine the efficacy and safety of first-line CC-486 plus CHOP in patients with Peripheral T-cell Lymphoma (PTCL) who have received no prior systemic therapy. The main objective is to determine the complete response rate (CR) of CC486-CHOP in PTCL. CR rate after cycle 6 will be used for the purpose of interim efficacy analysis.

* The study includes 6 cycles (~18 weeks) of treatment and 2 years of follow-up. The projected end date is 12/31/2022. Patients achieving complete remission will be evaluated every 6 months for 2 years or until disease progression. Patients who have disease progression will be contacted every 6 months to assess for survival status.
* Standard dose CHOP will be provided on day 1 of each cycle and repeat every 3 weeks for a total of 6 cycles.
* CC486 at 300 mg daily will be administered orally from day -6 to day 0 for cycle 1 priming, and on days 8-21 following cycles 1-5.
* Patients in CR/PR following 6 cycles of treatment have the option to proceed to consolidative autologous stem cell transplant.
* Will continue on treatment as long as they are responding to therapy and not experiencing unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

- Histologically confirmed diagnosis of PTCL of the following subtypes: Nodal T-cell lymphoma with T-follicular helper (TFH) phenotype (tumor cells must express 2 or 3 TFH-related antigens, including PD1, CD10, BCL6, CXCL13, ICOS, SAP and CCR5)* Angioimmunoblastic T-cell lymphoma Follicular T-cell lymphoma PTCL/NOS, T-follicular helper (TFH) variant PTCL-NOS Anaplastic large cell lymphoma, ALK negative Anaplastic large cell lymphoma, ALK positive with IPI > 2 Adult T-cell leukemia / lymphoma

* No prior systemic therapy for lymphoma
* Measurable disease defined by a tumor mass ≥ 1.5 cm in one dimension and measurable in two dimensions
* ECOG performance status ≤ 2

Exclusion Criteria:

* Known central nervous system (CNS) involvement by lymphoma
* Active viral infection with HIV or hepatitis type B or C (seropositive HBV patients are eligible if they are negative for HBV DNA by PCR and receive concomitant antiviral therapy).
* Prior history of malignancies other than PTCL unless the patient has been disease free for ≥ 5 years from the signing of the ICF.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2022-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jia Ruan, MD, Ph.D, Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medicine, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruan J, Moskowitz A, Mehta-Shah N, Sokol L, Chen Z, Kotlov N, Nos G, Sorokina M, Maksimov V, Sboner A, Sigouros M, van Besien K, Horwitz S, Rutherford SC, Mulvey E, Revuelta MV, Xiang J, Alonso A, Melnick A, Elemento O, Inghirami G, Leonard JP, Cerchietti L, Martin P. Multicenter phase 2 study of oral azacitidine (CC-486) plus CHOP as initial treatment for PTCL. Blood. 2023 May 4;141(18):2194-2205. doi: 10.1182/blood.2022018254. PMID 36796016
- [Derived] Yoon SE, Cho J, Kim YJ, Kim SJ, Kim WS. Real-World Efficacy of 5-Azacytidine as Salvage Chemotherapy for Angioimmunoblastic T-cell Lymphoma. Clin Lymphoma Myeloma Leuk. 2022 Nov;22(11):e972-e980. doi: 10.1016/j.clml.2022.07.009. Epub 2022 Jul 17. PMID 35995702

RESULTS

PARTICIPANT FLOW:
Groups:
- CC486 +CHOP: CC486 +CHOP
  CC-486 Administration: CC-486 at 300 mg once daily is to be administered Cycle 1, Day -6 to 0 and Cycles 1 to 5, Day 8 to 21. Antiemetic prophylaxis is recommended before dosing. All efforts should be made to administer CC-486 on all scheduled days of the Cycle 1 priming dosing (7 days, Cycle 1 Day -6 to Cycle 1 Day 0) and the Cycle 1-5 dosing (14 days, Day 8-21). A dose missed earlier in a day can be administered later that day as long as it is taken at least 8 hours before the next scheduled dose. Any missed dose should not be taken beyond the last scheduled day of CC-486 administration for the cycle, but should be returned by the subject for CC 486 accountability. If vomiting occurs after a dose of CC-486 is administrated, that dose should not be made up later that day.
  CHOP Administration: CHOP is to be administered on Days 1 to 5 of Cycles 1-6. Chemotherapy can be administer within +72h or -24h of Day 1 of each scheduled Cycle. Preparation and infusion rate are according to the package insert and local practice. The doses to be used are:
  Cyclophosphamide: 750 mg/m2 IV on day 1 Doxorubicin: 50 mg/m2 IV on day 1 Vincristine: 1.4 mg/m2 IV (not to exceed 2.0 mg total) on day 1 Prednisone: 100 mg PO days 1-5
Period: Treatment Phase
Arm/Group | CC486 +CHOP
Started | 21
Completed | 18
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1
Not completed — PD | 1
Period: Post-treatment Follow-up Phase
Arm/Group | CC486 +CHOP
Started | 15 (Three subjects did not enter follow-up: 1 had PD at EOT, 2 withdrew consent)
Completed | 0
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | CC486 +CHOP
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Description: Complete response rate (CR) of CC486-CHOP in PTCL by Lugano Criteria for target lesions, and the Deauville Criteria (5 point scale) assessed by PET or CT; CR (complete metabolic or radiologic response) defined as Deauville score of 1, 2 or 3 by PET or regression of all target lesions to < 1.5cm in longest diameter by CT.
Time Frame: After Cycle 6 at 18 weeks
Population: 3 of 21 participants did not complete treatment as outlined in the Participant Flow section; these subject were unevaluable and not included in analysis.
Measure: Number; unit: percentage of participants
Arm/Group | CC486 +CHOP
Number analyzed (Participants) | 18
percentage of participants | 75
Statistical Analysis 1: Comparison: CC486 +CHOP; Test type: Other; Proportion (percent) = 75.0, 95% CI 2-sided [46.5 to 90.3] — Exact (Clopper-Pearson) 95% confidence interval for complete response rate

2. Secondary Outcome: Kaplan-Meier Overall Survival
Description: Overall Survival (OS) assessed by Kaplan-Meier survival analysis. The Kaplan-Meier overall survival estimate at 2 years (with 95% confidence interval) is reported.
  OS defined as the time from first treatment day until death (or until last follow-up if alive).
Time Frame: 2 years
Population: 1 patient had missing overall survival information.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CC486 +CHOP
Number analyzed (Participants) | 20
percentage of participants | 68.0 [46.7 to 89.2]

3. Secondary Outcome: Kaplan-Meier Progression-Free Survival
Description: Progression-free survival (PFS) assessed by Kaplan-Meier survival analysis. The Kaplan-Meier progression-free survival estimate at 2 years (with 95% confidence interval) is reported.
  PFS defined as the time from first treatment day until objective or symptomatic progression or death (or date of last follow-up if no progression/death).
Time Frame: 2 years
Population: 1 participant had missing progression-free survival information.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CC486 +CHOP
Number analyzed (Participants) | 20
percentage of participants | 65.8 [43.4 to 88.1]

ADVERSE EVENTS:
Time Frame: From time of informed consent to 28 days post last dose of study drug, approximately 8 months.
Arm/Group | CC486 +CHOP
All-Cause Mortality (participants affected / at risk) | 1/21
Serious Adverse Events (participants affected / at risk) | 6/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC486 +CHOP (N=21)
Hyponatremia (Metabolism and nutrition disorders) | 1
Neutopenic Fever (Investigations) | 2
Diarrhea (Gastrointestinal disorders) | 1
Blood Bilirubin Increase (Metabolism and nutrition disorders) | 1
Stroke (Nervous system disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1
Influenza A (Infections and infestations) | 1
Headache (Nervous system disorders) | 1
Lung Infection, COVID-19 (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CC486 +CHOP (N=21)
Anemia (Blood and lymphatic system disorders) | 10
Sinus tachycardia (Cardiac disorders) | 3
Orthostatic hypotension (Cardiac disorders) | 3
Chest pain - cardiac (Cardiac disorders) | 3
Abdominal Pain (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 19
Diarrhea (Gastrointestinal disorders) | 11
Dry Mouth (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Mucositis Oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 15
Stomach Pain (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 10
Edema limbs (General disorders) | 6
Fatigue (General disorders) | 14
Fever (General disorders) | 3
Generalized weakness (General disorders) | 2
Non-cardiac chest pain (General disorders) | 4
Night sweats (General disorders) | 2
Weight loss (General disorders) | 2
Oral Candidiasis (Infections and infestations) | 2
Rhinovirus (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 13
Neutrophil count decreased (Investigations) | 15
Transaminitis (Investigations) | 2
Platelet count decreased (Investigations) | 11
White blood cell decreased (Investigations) | 12
Anorexia (Metabolism and nutrition disorders) | 6
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 6
Dysgeusia (Nervous system disorders) | 3
Headache (Nervous system disorders) | 5
Neuropathy (Nervous system disorders) | 5
Syncope (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 4
Insomnia (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 2
Superficial thrombophlebitis (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT03542266/Prot_SAP_000.pdf